CLINICAL TRIAL: NCT02627560
Title: The Effect of Topical Administration of Tranexamic Acid on Postoperative Bleeding and Seroma Formation in Patients Undergoing Mastectomy: A Prospective Placebo-controlled Double Blinded Randomized Study
Brief Title: The Effect of Topical Tranexamic Acid on Bleeding and Seroma Formation in After Undergoing Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015/1722; 2015-003160-37 (EudraCT Number)
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Hemorrhage; Breast Neoplasms; Seroma
Keywords: Administration, topical; Tranexamic acid; Postoperative care; Mastectomy
MeSH Terms: conditions — Postoperative Hemorrhage; Breast Neoplasms; Seroma | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical tranexamic acid (Experimental): tranexamic acid to be smeared on surgical wounds before closure
  Interventions: Drug: Tranexamic Acid
- placebo control (Placebo Comparator): saline to be smeared on surgical wounds before closure
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Tranexamic Acid — moisten the surgical wound surface with 20 ml tranexamic acid 25 mg/ml
  Arms: topical tranexamic acid
Drug: saline — moisten the surgical wound surface with 20 ml placebo (0.9% saline)
  Arms: placebo control

SUMMARY:
After surgical procedures, interventions to reduce postoperative bleeding are of great importance. In this study, the effect will be investigated of smearing tranexamic acid, which is designed for injection, directly onto the raw wound surface (topical application) created during surgery. Topical application allows a small amount of drug to reach a large wound area, higher drug concentration in the exposed wound surface but very low concentration in the body, and no risk of injury from needles. The researchers have recently shown that topically applicated tranexamic acid reduces bleeding in women who had two-sided breast reduction surgery. Now it will be studied whether topically applicated tranexamic acid reduces bleeding after breast surgery for breast cancer.

After surgery for breast cancer patients may also experience problems with long lasting seroma. Therefore it will at the same time be investigated whether topical tranexamic acid reduces the development of seroma in these patients.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* undergoing unilateral mastectomy with or without axillary node dissection
* received adequate oral and written information about the study and signed an informed-consent form

Exclusion Criteria:

* pregnant or breastfeeding
* known thromboembolic disease or with high risk of thromboembolism, warranting extra anticoagulation in connection with the procedure
* known allergy to tranexamic acid/Cyklokapron®

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
bleeding as defined by drain production per hour the first 24 hours | 24 hours postoperatively
  Drains are placed in surgical wounds during operation, and amount of blood on drains measured in ml

SECONDARY OUTCOMES:
Daily drain production up to drain removal - cumulative volume | 3 weeks
number of patients having surgical bleeding in need of re-operation | 3 weeks
number of postoperative aspirations of clinical seroma | up to 3 months
chronic seroma (lasting more than three months) | 3 months
  volume of seroma aspirated

CONTACTS AND LOCATIONS:
Overall Officials: Petter Aadahl, MD PhD, Study Director — St. Olavs Hospital; Sverrir Olafsson, Study Director — Ålesund Sykehus
Locations (2):
- Norway (2):
  - Department of Surgery, Aalesund Hospital, Ålesund
  - St Olavs University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843
- [Result] Ausen K, Hagen AI, Ostbyhaug HS, Olafsson S, Kvalsund BJ, Spigset O, Pleym H. Topical moistening of mastectomy wounds with diluted tranexamic acid to reduce bleeding: randomized clinical trial. BJS Open. 2020 Apr;4(2):216-224. doi: 10.1002/bjs5.50248. Epub 2019 Dec 26. PMID 32207575